CLINICAL TRIAL: NCT06241638
Title: Improving HbA1c Levels by Methylcobalamin Vitamin in Diabetic Volunteers, Combined With Dapagliflozin as Type Two Diabetes Mellitus Routine Treatment
Brief Title: Improving HbA1c Levels by Methylcobalamin Vitamin in Diabetic Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Balqa Applied University (Other)
Responsible Party: Principal Investigator, Walid Salem Aburayyan, Associate Professor, Al-Balqa Applied University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SREC-2022/783
Record Dates: First submitted 2024-01-18; First posted 2024-02-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vitamin B 12; dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin group (Active Comparator): Dapagliflozin group received only Dapagliflozin 10 mg/daily orally for twelve months
  Interventions: Drug: Dapagliflozin 10mg Tab
- Vitamin B12 and Dapagliflozin group (Experimental): Vitamin B12 and Dapagliflozin group received orally Vit. B12 supplements methylcobalamin 500 µg once daily with their usual anti-diabetic therapy Dapagliflozin 10 mg/daily for twelve months.
  Interventions: Drug: Vitamin B12 0.5 MG/ACTUAT; Drug: Dapagliflozin 10mg Tab

INTERVENTIONS:
Drug: Vitamin B12 0.5 MG/ACTUAT — The investigators measured the blood levels of Vitamin B12 and HbA1c as well as the BMI in two study groups; The Experimental group: Vitamin B12 and Dapagliflozin group and Active Comparator group: Dapagliflozin group.
  The Dapagliflozin group received only Dapagliflozin 10 mg/daily orally for twelve months, whereas, the Vitamin B12 and Dapagliflozin group received Vit. B12 supplements methylcobalamin 500 µg once daily orally with the anti-diabetic therapy Dapagliflozin 10 mg/daily orally for twelve months.
  Arms: Vitamin B12 and Dapagliflozin group
Drug: Dapagliflozin 10mg Tab — The investigators measured the blood levels of Vitamin B12 and HbA1c as well as the BMI in two study groups; The Experimental group: Vitamin B12 and Dapagliflozin group and Active Comparator group: Dapagliflozin group.
  The Dapagliflozin group received only Dapagliflozin 10 mg/daily orally for twelve months, whereas, the Vitamin B12 and Dapagliflozin group received Vit. B12 supplements methylcobalamin 500 µg once daily orally with the anti-diabetic therapy Dapagliflozin 10 mg/daily orally for twelve months.

SUMMARY:
The current study was conducted to evaluate the prognostic implications of vitamin B12 admission on BMI and HbA1c levels in type 2 diabetic patients treated with Dapagliflozin as a routine medication.

DETAILED DESCRIPTION:
Eighty diabetic patients were enrolled in this study; 37 females and 43 males with inclusion criteria of vitamin B12 levels less than 233 ng/ml. The participants were divided into two groups, the Dapagliflozin group (active comparator group) received only the diabetic-controlling drug Dapagliflozin 10 mg/daily orally for twelve months, whereas, vitamin B12 and Dapagliflozin group (Experimental group) received Vit. B12 supplements as methylcobalamin 500 µg orally once daily with Dapagliflozin 10 mg/daily orally for twelve months. Glycemic control was measured by monitoring levels of HbA1c and Vitamin B12 in the participant's blood four times at time intervals of three months during the study period. Additionally, the weight measurements were recorded during the study period at time intervals of three months and BMI was calculated. The data obtained was treated by statistical analysis using SPSS software (version 20) for the significant correlation of the independent variables of the study groups after vitamin B12 supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patient treated with Dapagliflozin

Exclusion Criteria:

* The levels of Vitamin B12 more than 200 ng/ml

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
HbA1c in the two groups | One year
  The diabetic status in the two groups was evaluated by measuring the HbA1c levels

CONTACTS AND LOCATIONS:
Locations (1):
- Walid Aburayyan, Salt, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aburayyan W, Zakaraya Z, Hamad M, Majali IS, Abu Dayyih W, Seder N, Alkhadeir H, Khaleel A. Improving HbA1c Levels by Methylcobalamin Vitamin in Diabetic Volunteers, Combined with Dapagliflozin as Type 2 Diabetes Mellitus Routine Treatment: A Controlled Randomized, Double-blind Trial. Iran J Med Sci. 2025 May 1;50(5):324-333. doi: 10.30476/ijms.2024.101606.3423. eCollection 2025 May. PMID 40433181